CLINICAL TRIAL: NCT03839953
Title: Exercise Rehabilitation for Critical Limb Ischemia Patients After Revascularization: Pilot Randomized Controlled Trial Assessing Functional Capacity and Quality of Life After a 12-week Rehabilitation Program Versus Best Medical Therapy
Brief Title: Exercise Rehabilitation for Patients With Critical Limb Ischemia After Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Randy Moore, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB17-730
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
Keywords: Rehabilitation; Exercise; Revascularization; Endovascular; Vascular Surgery
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Medical Therapy (Active Comparator): After undergoing revascularization for critical limb ischemia, patients will receive best medical therapy under the supervision of a vascular internal medicine specialist. This care will include advice on smoking cessation, physical activity guidelines, blood pressure regulation, statin administration and possible anti-platelet administration.
  Interventions: Other: Best Medical Therapy
- Supervised Exercise Program (Experimental): Patients will receive best medical therapy plus participation in a 12-week supervised exercise program.
  Interventions: Behavioral: Supervised Exercise Program

INTERVENTIONS:
Behavioral: Supervised Exercise Program — This intervention is a 12-week supervised exercise program at an established cardiac rehabilitation facility.
  Arms: Supervised Exercise Program
Other: Best Medical Therapy — After undergoing revascularization for critical limb ischemia, patients will receive best medical therapy under the supervision of a vascular internal medicine specialist. This care will include advice on smoking cessation, physical activity guidelines, blood pressure regulation, statin administration and possible anti-platelet administration.
  Arms: Best Medical Therapy

SUMMARY:
Peripheral arterial disease (PAD) affects more than 200 million people worldwide. This disease occurs with narrowing and occlusion of arteries supplying oxygenated blood to the organs and limbs. Symptomatic patients typically experience leg pain with physical activity. More advanced disease states are referred to as critical limb ischemia (CLI), where patients may have leg pain at rest or non-healing wounds. Primary treatment of PAD involves risk factor management; smoking cessation, management of blood pressure, blood cholesterol, diabetes, and exercise prescription. Patients with CLI typically require interventions to reestablish blood supply to their limbs. There is currently minimal understanding of the role for exercise rehabilitation after revascularization procedures in this vulnerable population. This is the first clinical to understand the role of exercise for these patients. We hypothesize that exercise rehabilitation after revascularization will improve quality of life and functional capacity in these patients.

DETAILED DESCRIPTION:
Background: Peripheral arterial disease (PAD) refers to narrowing and occlusion of arteries supplying oxygenated blood to non-coronary and non-intracranial circulatory systems. This term is typically used to describe disease in the legs though it also affects upper extremities, renal and mesenteric vessels. Symptomatic patients typically experience leg pain with walking or physical activity which is referred to as intermittent claudication (IC). In more advanced chronic disease states with severely compromised blood flow to the tissues, patients may have leg pain at rest or even non healing wounds that can lead to tissue loss which is defined as critical limb ischemia (CLI).

Risk factor management is critical for PAD patients with the goal of improving symptoms and preventing disease progression. This includes smoking cessation as well as appropriate management for hypertension, dyslipidemia and diabetes. Antiplatelet therapy should be initiated in symptomatic patient or when other risk factors are present. Exercise interventions should be encouraged in all patients with PAD. In patients who have progressed to critical limb ischemia, treatment goals are to relieve pain, heal wounds and prevent limb loss. In addition to risk factor management and medical therapy, these patients require revascularization procedures. Depending on the extent and location of disease, the techniques used may be endovascular/interventional (minimally invasive), surgical, or a hybrid combination of the two.

There has been minimal research examining exercise rehabilitation after revascularization. There are no studies that have focused on exercise rehabilitation exclusively in patients with CLI.

Purpose/Objectives: The aim of this study is to develop a better understanding of the role for supervised exercise rehabilitation programs (SEP) in PAD-CLI patients after revascularization. This pilot study will assess the feasibility for expanding this research to a larger randomized controlled trial.

Study Design:

This is a two-phase, single-center, non-blinded randomized controlled trial.

Objectives:

In phase 1, the investigators will assess feasibility. Specifically, the investigators will assess rate of enrollment, barriers to participation and any methodological challenges that may require changes. If phase 1 of this study shows reasonable rates of enrollment and no methodological challenges, we will proceed to phase 2.

Key objectives for phase 2 are as follows:

1. The primary objective is to show how SEP affects functional capacity and quality of life in patients with PAD-CLI after revascularization.
2. The secondary objective is to show how SEP affects the rate of major adverse limb events (MALE) and improve survival in patients with PAD-CLI after revascularization.

Hypotheses: 1) PAD-CLI patients who have undergone revascularization will have a greater improvement in functional capacity and quality of life compared with patients treated with best medical therapy alone.

2) PAD-CLI patients who have undergone revascularization will have fewer MALE and improved survival compared with patients treated with best medical therapy alone.

Methodology: Patients included in the study will be identified in the vascular surgery outpatient clinic or through emergency department as requiring revascularization secondary to critical limb ischemia. Patients will be approached regarding study participation prior to the revascularization procedure. After eligibility is confirmed and patients have signed informed consent, patients will be randomized to one of two groups:

1. Best Medical Therapy (BMT): Appropriate risk factor management, encouragement to mobilize.
2. Supervised Exercise Program (SEP): consist of BMT plus a supervised exercise program.

Patients will undergo evaluation of functional capacity assessment using a graded treadmill test at the outset of the study and after 12 weeks of either BMP or SEP. The investigators will also administer a validated quality of life (QoL) questionnaire to the two different groups at the outset and completion of the study. Patients will be followed annually to monitor for MALE and survival.

Statistics: Normally distributed data will be presented as mean ± SD. Results at baseline and 12 weeks will be compared using a paired t-test. For data that is not normally distributed, comparisons will be performed using a non-parametric Mann-Whitney test. Comparisons will be accepted as statistically significant at 95% confidence level (p≤0.05). STATA software will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulating prior to procedure
2. Living independently prior to procedure
3. Available to attend all SEP and follow-up appointments
4. PAD Fontaine class III and IV (rest pain and tissue loss)
5. Entry with consent of vascular surgeon
6. Ischemia secondary to TASC A-D lesions identified on imaging (CTA or angiogram)
7. Able to understand and sign informed consent
8. >18 years of age

Exclusion Criteria:

1. Confined to wheelchair
2. Patients with exercise tolerance limitations due to other co-morbidities such as cardiorespiratory, musculoskeletal, or peripheral neuropathy. (NYHA class III and IV)
3. PAD Fontaine class I and II (asymptomatic, claudication)
4. Patients with ongoing tissue loss that limits ambulation
5. Patient with previous revascularization procedures
6. Patients undergoing revascularization for acute limb ischemia events

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of enrollment | 3 months
  A minimum of 3 patients per month should be enrolled
Functional Capacity | Three months
  Functional capacity will be evaluated by a six-minute walk test
Quality of Life assessed by VascuQuol questionnaire | Three months
  Questionnaire with 25 items validated for patients with peripheral arterial disease
Health status assess by SF-36 | Three months
  36-item self-reported survey that provides a measure of patient health
Barriers or experiences with physical activity | Three months
  We will conduct a 30-minute interview to gain better understanding of patient experiences with exercise rehabilitation.

SECONDARY OUTCOMES:
Major adverse limb events (MALE) | Five years
  Clinical deterioration or condition requiring surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Moore, MD, Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Center, Alberta Health Services, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT03839953/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT03839953/ICF_001.pdf